CLINICAL TRIAL: NCT06595589
Title: The Effect of Dental Caries Conceptualizing and the Residential University Life on the Caries Prevalence and Caries Prevention Practice of Egyptian Dental Students: Observational Cross-Sectional Study.
Brief Title: Effect of Caries Conceptualizing and Residential University Life
Status: Not yet recruiting | Type: Observational
Sponsor: Sara Ibrahim Ahmed Hedia (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Sara Ibrahim Ahmed Hedia, Teaching Assistant in conservative department at Galala University, Cairo University
Organization: Cairo University (Other)
Other Study IDs: Conceptualization of Caries
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Caries, Dental
Keywords: caries prevalence; residential students; dental students
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to detect the conceptualization of dental caries among dental student and compare the caries prevalence in residential and non residential dental student

DETAILED DESCRIPTION:
A face-to-face meeting will be held with the target student group, illustrating the study set up and seeking the participation approval. The students who will accept to participate in the study will receive a questionnaire including the caries conceptualization assessment inquiry, the caries prevention practice as well as the residential habits. All the participating students will be scheduled for dental examination to record their DMFT index. The digital responses will be coded, analyzed and correlated with the clinical findings.

ELIGIBILITY:
Inclusion criteria will be:

* Students already taught a dental cariology in 4th year of university.
* Students registered in the Galala dental program science year one.
* Medically free students.
* Students having at least 1year clinical practice.

Exclusion criteria will be:

* First, second-, and third-year students.
* Non dental students.

Ages: 20 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young Adult 4th year Dental students
Sampling Method: Non-Probability Sample
Enrollment: 303 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Caries Prevalence | At base line Immediately after collecting the data
  DMFT (Decay, Missed, Filled teeth) index developed by World Health Organization (WHO) using numbered scores. (higher scores mean a worse outcome).
  Oral and dental examination were performed using a prob, mirror, and cotton rolls, in order to score each participant using DMFT index.

SECONDARY OUTCOMES:
caries conceptualization in relation to the Caries preventive behavior of the students. | At base line
  Scores (C1:C6) Questionnaire